CLINICAL TRIAL: NCT05113355
Title: Chidamide and Sintilimab for Chemotherapy-refractory Advanced High-grade Neuroendocrine Neoplasm: a Prospective, Single-arm, Multicenter, Phase 2 Clinical Study
Brief Title: Chidamide Plus Sintilimab for Chemotherapy-refractory Advanced High-grade Neuroendocrine Neoplasm
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other); Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-3197D
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Tumor Grade 3; Neuroendocrine Carcinoma; Neuroendocrine Neoplasm
Keywords: Histone Deacetylase Inhibitors; Chidamide; Neuroendocrine Neoplasm; PD-1; Sintilimab
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide + Sintilimab (Experimental): Experimental arm will be treated by chidamide combined with sintilimab for up to 24 months.
  Interventions: Drug: Chidamide; Drug: Sintilimab

INTERVENTIONS:
Drug: Chidamide — 30mg; administered orally; twice a week (d1, d4, d8, d11, d15, d18). Repeat every 3 weeks for up to 24 months.
  Other Names: Epidaza
Drug: Sintilimab — 200mg; intravenous infusion; d1. Repeat every 3 weeks for up to 24 months.
  Other Names: Tyvyt

SUMMARY:
The purpose of this study is to explore the efficacy and safety of chidamide combined with sintilimab in chemotherapy-refractory advanced high-grade neuroendocrine neoplasm.

DETAILED DESCRIPTION:
This study is a single-arm, multi-center, two-stage, phase II clinical trial conducted in China. This study adopts Simon's two-stage design, and the inclusion criteria and exclusion criteria of the two stages were consistent. Six patients with high-grade neuroendocrine neoplasm will be enrolled in the first stage. If more than one complete or partial responses were seen at planned interim analysis, the additional 17 patients will be recruited in the second stage and a total of 23 patients will be treated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Histologically confirmed advanced and metastatic high-grade neuroendocrine neoplasm;
3. Receive ≤ 2 types of chemotherapy for high-grade neuroendocrine tumors and had tumor progression;
4. ECOG ≤ 2;
5. Have at least one measurable lesion according to RECIST version 1.1;
6. Absolute neutrophil count ≥ 1.5×109 / L, platelet count ≥ 100×109 / L, hemoglobin ≥ 90 g/L;
7. Provide tumor samples for pathological diagnosis and PD-L1 biomarker detection;
8. Have ability to sign a written informed consent.

Exclusion Criteria:

1. Small cell lung cancer;
2. Have surgery or trauma within 4 weeks before enrollment, or are expected to receive surgical treatment;
3. Previous use of HDAC inhibitors;
4. Previous use of PD-1/PD-L1/PD-L2/CTLA-4 inhibitors;
5. Allergy to related drug components;
6. Have a medical history of immune deficiency diseases, or organ transplantation;
7. Have active autoimmune diseases requiring treatment or a medical history of autoimmune diseases in the past 2 years;
8. Have uncontrolled or significant cardiovascular disease;
9. Abnormal liver function (total bilirubin > 1.5×upper limit of normal); Transaminases (ALT/AST) >2.5×upper limit of normal (>5x upper limit of normal for patients with liver metastases), abnormal renal function (serum creatinine > 1.5×upper limit of normal);
10. Pregnancy ;
11. Receive any live or live attenuated vaccine within 4 weeks before enrollment;
12. Have serious diseases that may endanger the safety of patients, or affect patients to complete the research;
13. Any serious mental or cognitive disorder;
14. Patients are currently enrolled in another drug clinical trial within 4 weeks prior to enrollment;
15. Any other condition which is inappropriate for the study in the opinion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  Percentage of participants with complete response and partial response, assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 2 years
  Percentage of participants with complete response, partial response, and stable disease assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
Progression-free Survival (PFS) | Time from the date of enrollment to the earliest of documented disease progression or death, assessed up to 2 years
  Time from the date of enrollment until progression or death, whichever is first met
Overall Survival (OS) | Time from the date of enrollment to the earliest of documented death, assessed up to 3 years
  Time from the date of enrollment until death
Treatment-related Adverse Events (Safety) | Up to 2 years
  Frequency and grade of adverse events (the grade of adverse events is assessed according to CTCAE v4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Chunmei Bai, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not available to others.